CLINICAL TRIAL: NCT00030745
Title: Preoperative Chemotherapy Of Potentially Resectable Mesothelioma Of The Pleura
Brief Title: Combination Chemotherapy Before Surgery in Treating Patients With Mesothelioma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 17/00; SWS-SAKK-17-00 (Other: SAKK); EU-20136
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Malignant Mesothelioma
Keywords: stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have mesothelioma of the lung.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the proportion of patients with potentially resectable mesothelioma of the pleura remaining operable after treatment with neoadjuvant cisplatin and gemcitabine.
* Determine the response rate and overall survival of patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Determine the number of postoperative hospitalization days and occurrence and duration of surgical complications in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Compare the proportion of patients who report psychological distress at 3 months after surgery vs at study registration.

OUTLINE: Patients receive cisplatin IV on day 1 and gemcitabine IV on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses. Within 6 weeks after completion of chemotherapy, patients undergo restaging by CT scan followed by surgical resection.

Quality of life is assessed at baseline, day 1 of course 3, within 4 weeks after surgery, and then at 3 and 6 months.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 61 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and clinically confirmed pleural mesothelioma

  * Stages T1-3, N0-2, M0 by CT scan of the chest

    * Mediastinoscopy required for staging of mediastinal lymph nodes
  * Considered completely resectable

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No severe liver disease

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiac:

* Adequate cardiac function
* No cardiac disease that would preclude forced hydration or surgery

Pulmonary:

* Predicted postoperative FEV_1 greater than 1 by spirometry

Other:

* No contraindication to surgery
* No other prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No uncontrolled infection
* No uncontrolled diabetes
* No neurologic or psychiatric disorders that would preclude study compliance
* No other serious illnesses that would preclude study participation
* No other circumstances that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior pleurectomy or lung resection except for diagnostic purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2000-06; Primary Completion 2003-05 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf A. Stahel, MD, Study Chair — UniversitaetsSpital Zuerich
Locations (1):
- UniversitaetsSpital, Zurich, Switzerland

REFERENCES:
- [Result] Weder W, Stahel RA, Bernhard J, Bodis S, Vogt P, Ballabeni P, Lardinois D, Betticher D, Schmid R, Stupp R, Ris HB, Jermann M, Mingrone W, Roth AD, Spiliopoulos A; Swiss Group for Clinical Cancer Research. Multicenter trial of neo-adjuvant chemotherapy followed by extrapleural pneumonectomy in malignant pleural mesothelioma. Ann Oncol. 2007 Jul;18(7):1196-202. doi: 10.1093/annonc/mdm093. Epub 2007 Apr 11. PMID 17429100